CLINICAL TRIAL: NCT03739944
Title: Randomized Trial of Different Surgical Approaches in Patients of Chinese Early-stage Cervical Cancer
Brief Title: Different Surgical Approaches in Patients of Early-stage Cervical Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RACC
Record Dates: First submitted 2018-11-08; First posted 2018-11-14 (Actual); Last update posted 2018-12-28 (Actual); Status verified 2018-12

CONDITIONS: Uterine Cervical Neoplasm; Laparotomy; Laparoscopy; Survival; Mortality; Morbidity; Quality of Life; Pelvic Floor Disorders; Cost-Benefit Analysis
MeSH Terms: conditions — Uterine Cervical Neoplasms; Pelvic Floor Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Laparotomic radical hysterectomy (Active Comparator)
  Interventions: Procedure: Laparotomic radical hysterectomy
- Laparotomic radical trachelectomy (Active Comparator)
  Interventions: Procedure: Laparotomic radical trachelectomy
- Laparoscopic radical hysterectomy (Active Comparator)
  Interventions: Procedure: Laparoscopic radical hysterectomy
- Laparoscopic radical trachelectomy (Active Comparator)
  Interventions: Procedure: Laparoscopic radical trachelectomy

INTERVENTIONS:
Procedure: Laparotomic radical hysterectomy — Laparotomic radical hysterectomy for patients without fertility requirement
  Arms: Laparotomic radical hysterectomy
Procedure: Laparotomic radical trachelectomy — Laparotomic radical hysterectomy for patients with fertility requirement
  Arms: Laparotomic radical trachelectomy
Procedure: Laparoscopic radical hysterectomy — Laparoscopic radical hysterectomy for patients without fertility requirement
  Arms: Laparoscopic radical hysterectomy
Procedure: Laparoscopic radical trachelectomy — Laparoscopic radical hysterectomy for patients with fertility requirement
  Arms: Laparoscopic radical trachelectomy

SUMMARY:
This multi-center, randomized controlled study aims to compare the survival outcomes (including overall survival, progression-free survival and disease-free survival between Chinese uterine cervical patients receiving different surgical routes (laparotomy and laparoscopy) for radical hysterectomy or trachelectomy, which is the primary study objective. All patients with uterine cervical cancer of FIGO stage IA1 (with lymphovascular space invasion), IA2 and IB1 will be included and randomized into two groups: laparotomy and laparoscopy groups for radical hysterectomy or trachelectomy. Secondary study objectives include: patterns of recurrence, treatment-associated morbidity (6 months from surgery), cost-effectiveness, pelvic floor function, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed primary adenocarcinoma, squamous cell carcinoma or adenosquamous carcinoma of the uterine cervix
* FIGO stage IA1 (with lymphovascular space invasion), IA2 or IB1
* Type II or III radical hysterectomy or trachelectomy
* Performance status of ECOG 0-1
* Aged 18 years or older
* Signed an approved informed consents

Exclusion Criteria:

* Not satisfying any of the inclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2018-11-23 (Actual); Primary Completion 2022-11-23 (Estimated); Study Completion 2023-11-23 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Five years
  The length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse.

SECONDARY OUTCOMES:
Overall survival | Five years
  The length of time from either the date of diagnosis or the start of treatment for a disease, such as cancer, that patients diagnosed with the disease are still alive.
Disease-free survival | Five years
  In cancer, the length of time after primary treatment for a cancer ends that the patient survives without any signs or symptoms of that cancer.
Morbidity rate | Six months
  Refers to having a disease or a symptom of disease, or to the amount of disease within a population. In this study, morbidity of six months from the surgery is defined according to Common Terminology Criteria for Adverse Events (CTCAE) v4.03

OTHER OUTCOMES:
Cost-effectiveness of different surgical routes | One year
  The direct cost of different surgical routes
Quality of life | Three years
  The quality of life measured by academic questionnaire
Sex function | Five years
  Sex function measured by academic questionnaire before and after surgeries
Urodynamics | Five years
  Urinary functions are measured by dynamic tests before and after surgeries
Rectal functions | Five years
  Rectal functions are measured by dynamic tests before and after surgeries

CONTACTS AND LOCATIONS:
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The data will be available to all the researches via public websites.
Supporting Information: Study Protocol, CSR
Time Frame: The data will be available once the papers were accepted and be available for ever

REFERENCES:
- [Derived] Chao X, Li L, Wu M, Wu H, Ma S, Tan X, Zhong S, Lang J. Minimally invasive versus open radical trachelectomy for early-stage cervical cancer: protocol for a multicenter randomized controlled trial in China. Trials. 2020 Dec 14;21(1):1022. doi: 10.1186/s13063-020-04938-3. PMID 33317612
- [Derived] Ferrandina G, Corrado G, Scambia G. Minimally invasive surgery and quality of life in cervical cancer. Lancet Oncol. 2020 Jun;21(6):746-748. doi: 10.1016/S1470-2045(20)30161-3. No abstract available. PMID 32502439
- [Derived] Chao X, Li L, Wu M, Ma S, Tan X, Zhong S, Lang J, Cheng A, Li W. Efficacy of different surgical approaches in the clinical and survival outcomes of patients with early-stage cervical cancer: protocol of a phase III multicentre randomised controlled trial in China. BMJ Open. 2019 Jul 29;9(7):e029055. doi: 10.1136/bmjopen-2019-029055. PMID 31362966